CLINICAL TRIAL: NCT05135455
Title: VAXZEVRIA Intramuscular Injection General Use Result Study for the Long-term Safety of VAXZEVRIA
Brief Title: VAXZEVRIA Japan Post-Marketing Surveillance (PMS) for the Long-term Safety of VAXZEVRIA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8111C00005
Record Dates: First submitted 2021-11-16; First posted 2021-11-26 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Prevention of Infectious Disease Caused by SARS-CoV-2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
This survey will be conducted for the subjects who participate in the priority survey (cohort survey) conducted by the Scientific Research Group of the Ministry of Health, Labour and Welfare at the initial stage of administration of the COVID-19 vaccination. The present study aims to collect information on serious adverse events or COVID-19 infection observed from 28 days after the last vaccination of VAXZEVRIA up to 12 months after the last vaccination and to evaluate the long-term safety of this vaccine.

DETAILED DESCRIPTION:
This survey will be conducted for the subjects who participate in the priority survey (cohort survey) conducted by the Scientific Research Group of the Ministry of Health, Labour and Welfare at the initial stage of administration of the COVID-19 vaccination.

The present study aims to collect information on serious adverse events (including Thrombosis in combination with thrombocytopenia, Immune-mediated neurological conditions, Vaccine-associated enhanced disease (VAED) including Vaccine-associated enhanced respiratory disease(VAERD), Thrombosis or other diseases) or COVID-19 infection observed from 28 days after the last vaccination of VAXZEVRIA up to 12 months after the last vaccination and to evaluate the long-term safety of this vaccine.

ELIGIBILITY:
Inclusion Criteria:

The subjects who participated in the cohort study conducted by the Scientific Research Group of the MHLW and those who give written consents for this study.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects who participated in the cohort study conducted by the Scientific Research Group of the MHLW and those who give written consents for this study.
Sampling Method: Non-Probability Sample
Enrollment: 467 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
The incidence of SAEs will be calculated by preferred term (PT) by overall and with/without causal relationships with VAXZEVRIA assessed by investigator(s). | From the next day of 28 days after the last vaccination of VAXZEVRIA up to 12 months after the last vaccination.
  The incidence of SAEs (including thrombosis in combination with thrombocytopenia, immune-mediated neurological conditions and VAED including VAERD, thrombosis or other diseases) will be calculated by preferred term (PT) by overall and with/without causal relationships with VAXZEVRIA assessed by investigator(s).
Number of the subjects considered to be severe case of COVID-19 and its incidence (%) will be calculated. The subject who required a hospitalization in intensive care unit or use of respirator will be defined as a severe case. | From the next day of 28 days after the last vaccination of VAXZEVRIA up to 12 months after the last vaccination.
  Number of the subjects considered to be severe case of COVID-19 and its incidence (%) will be calculated. The subject who required a hospitalization in intensive care unit or use of respirator will be defined as a severe case based on the severity classification reference of "A guide for front-line healthcare workers (MHLW, 2020)". Ad hoc analysis might be performed as necessary.

CONTACTS AND LOCATIONS:
Locations (6):
- Japan (6):
  - Research Site, Chiba
  - Research Site, Hyōgo
  - Research Site, Kumamoto
  - Research Site, Mie
  - Research Site, Shizuoka
  - Research Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR Synopsis for D8111C00005 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8111C00005&attachmentIdentifier=aaf6bbf9-16cb-454a-90e9-48d547eb9c75&fileName=Redacted_CSR_Synopsis_for_D8111C00005.pdf&versionIdentifier=